CLINICAL TRIAL: NCT04889352
Title: Optimizing Timing of Follow-up Colonoscopy: A Pilot Cluster Randomized Trial to Test the Utility of a Knowledge Translation Tool
Brief Title: Optimizing Timing of Follow-up Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2020:435
Record Dates: First submitted 2021-04-15; First posted 2021-05-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Colo-rectal Cancer; Colon Polyp; Colonic Polyp; Rectal Polyp; Polyp of Colon; Polyp Rectal; Polyps
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Polyps

STUDY DESIGN:
Intervention Model Description: This will be a cluster randomized controlled trial in which individual endoscopy physicians (gastroenterologists and surgeons) will be randomized (stratified by physician specialty) to one of two groups: A) provided access to the application (intervention group) or B) not provided access to the application (control group). The clusters of patients will be defined by the endoscopy physician providing the colonoscopy.
Who Masked: Investigator
Masking Description: Randomization will be performed after the endoscopy physician consent and enrolment into the study. A computer generated randomization sequence will used in blocks of eight. Stratification for surgical and gastroenterology endoscopy physician will be performed as there might be differential adherence to recommendations by specialty of training.Randomization will be performed and the application distributed by study personnel different than those involved in data extraction from medical records so that the person extracting the data remains blinded to the randomized group assignment. Patients of participating physicians will not require blinding as they will not be approached by the study investigators and will get routine care decided by their physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Access to colonoscopy web app (Experimental): Approximately half of the consenting individual endoscopy physicians in the city (gastroenterologists and surgeons) will be randomized (stratified by physician specialty) to the intervention group where they are provided access to an application which indicates recommended timing of follow-up colonoscopy given values for various entered factors. In the intervention group, the application can be downloaded to smart phones for portability which will allow access in an endoscopy suite or in clinic or used as a reference at other times. It can also be accessed online (all endoscopy rooms in Winnipeg have computers with internet access for the endoscopy physicians' use). Access to the application will be password-protected, thereby avoiding exposure of the non-intervention group to the application. The clusters of patients will be defined by the endoscopy physician providing the colonoscopy.
  Interventions: Other: Access to colonoscopy web app
- Control (No Intervention): Approximately half of the consenting individual endoscopy physicians in the city (gastroenterologists and surgeons) will be randomized (stratified by physician specialty) to the group where they are not provided access to the application (control group).

INTERVENTIONS:
Other: Access to colonoscopy web app — There is a very high utilization of colonoscopy at both shorter and longer time intervals than the recommended guidelines. Investigators have developed a clinical support tool in which the characteristics of the patients can be inputted and the guideline recommended time interval for surveillance colonoscopy is then provided. This tool uses the recommendations from the current North American national guidelines. The tool has been developed as a web-based application as well as a smart phone application.
  Arms: Access to colonoscopy web app

SUMMARY:
Overall Objective: To optimize timing of surveillance colonoscopy.

Principal research question and specific aims: To assess the impact of access to a hand-held application on the timing of surveillance colonoscopy. To assess whether access to the tool improves adherence to recommended guidelines for follow-up colonoscopy intervals.

Colonoscopy is commonly used for surveillance of patients with high risk of developing colorectal cancer, including those with family history of colorectal cancer and those with colorectal polyps. The recommended timing of surveillance colonoscopy varies by the estimated risk for development of colorectal cancer. The estimated risk varies by family history of colorectal cancer (number of affected individuals, age of the persons affected with CRC) and characteristics of the colorectal polyps (size, number, and histology of colorectal polyps (tubular or villous; high grade or low-grade dysplasia; sessile serrated polyp, sessile serrated polyp with dysplasia, hyperplastic polyp or traditional serrated adenomas). Guidelines take all of these factors into account in the recommendations for follow-up colonoscopy and hence are difficult to recall for the busy clinicians. Colonoscopy surveillance is frequently performed at shorter or longer than the recommended time intervals. The investigators have developed a smart phone application in which the characteristics of the patients can be inputted and the tool provides the recommended time interval for surveillance colonoscopy, based on North American guidelines. The investigators are proposing a pilot randomized trial to determine sample size estimates for a larger trial to assess the utility of this application in clinical practice.

DETAILED DESCRIPTION:
Study design and intervention: This will be a cluster randomized controlled trial in which individual endoscopy physicians (gastroenterologists and surgeons) will be randomized (stratified by physician specialty) to one of two groups: A) provided access to the application (intervention group) or B) not provided access to the application (control group). In the intervention group, the application can be downloaded to smart phones for portability which will allow access in an endoscopy suite or in clinic or used as a reference at other times. It can also be accessed online (all endoscopy rooms in Winnipeg have computers with internet access for the endoscopy physicians' use). The clusters of patients will be defined by the endoscopy physician providing the colonoscopy.

Intervention: Access to the application which will be available both as a web-based as well as a smart phone application.

Setting: Colonoscopies included in the study will be those performed in the Winnipeg endoscopy units.

A research assistant will extract data from medical records maintained by the hospitals and physicians privately. Individual cases of colonoscopies will be identified through the city-wide endoscopy program database. Study data will be collected and managed using the REDCap (Research Electronic Data Capture) electronic data capture tools hosted at the University of Manitoba.

Concealment of Allocation and Randomization: Randomization will be performed after the endoscopy physician consent and enrollment into the study. A computer generated randomization sequence will used in blocks of eight. Stratification for surgical and gastroenterology endoscopy physician will be performed as there might be differential adherence to recommendations by speciality of training.

Blinding: Randomization will be performed and the application distributed by study personnel different than those involved in data extraction from medical records so that the person extracting the data remains blinded to the randomized group assignment.

Patient consent: Patients will not be approached by the study investigators and will get routine care decided by their physicians. Information on recommendations will be extracted from medical records retrospectively; hence, patient consent will not be required.

Duration of treatment and duration of follow-up: This is a cross-sectional study of those undergoing colonoscopy with no follow-up after any pathology is reported.

Outcomes: The primary outcome of analysis will be congruence (agreement) of the colonoscopy physician recommendation with the guideline recommendation.

Endoscopy physician recommendations will be determined from review of the medical records (endoscopy reports and letters/notes in the medical charts). Listing of colonoscopies performed by each enrolled colonoscopy physician will be obtained from the centralised common endoscopy reporting system. Absence of documented recommendations will be considered an incongruent recommendation in the primary analysis and excluded in a sensitivity analysis.

Medical records will be reviewed to obtain the history relevant to determining the timing of surveillance (characteristics of polyps, family history, inclusion and exclusion criteria). Absence of documented relevant history will be considered an incongruent recommendation in the primary analysis and excluded in a sensitivity analysis.

Secondary outcomes will be collected by a survey distributed to the group of endoscopy physicians that were provided the app to determine their opinions about the app. The survey will inquire about ease of use, perception of reliability, likelihood of future use, whether the app provided helpful information and how often they used the app and when. Percentage responses will be tabulated for this descriptive outcome. Investigators will also include open-ended questions about any desired changes to the app.

Another secondary outcome will be the proportion of cases which have a documented recommendation.

Similarly, in this pilot study, the investigators will assess the proportion of the medical records which have complete information (family history of colorectal cancer/polyps, different polyp characteristics) required to make surveillance colonoscopy recommendations as per the guidelines.

ELIGIBILITY:
Inclusion Criteria:

For physician participants, there are no age limits/parameters. All physicians performing colonoscopy on adult patients in Winnipeg will be eligible to participate (other than those involved in pilot testing and study investigators). Participating physicians will be informed that the introduced intervention will be an information tool to help improve care for individuals undergoing colonoscopy, and will be asked to consent to review of their patient records. Participating physicians will be informed that no individual-level information will be disclosed at any time and all analysis will be on anonymized data.

For patient participants:

* Patients must be older than 50 years and up to 75 years old for inclusion in the study data.
* Adequate bowel preparation defined by Boston Bowel Preparation Scale Score of ≥ 2 in each of segments of the colon (Boston bowel prep scale score recording is mandatory in the Winnipeg city-wide endoscopy reporting system);
* Colonoscopy completed to the cecum/ileocolonic anastomosis;
* Colonoscopy performed between 1 to 4 months before randomization of endoscopy physician (to determine baseline adherence) or between 3 to 7 months after randomization (to determine effect of the intervention).

Exclusion Criteria:

Physicians will be excluded if they are away for more than six weeks continuously in the six months after randomization. In this situation, an alternate physician will be recruited and randomized. Thus there is no anticipated loss of follow-up.

Patients will be excluded if any of the following criteria are met:

1. History of inherited CRC predisposition (Lynch Syndrome, Familial adenomatous polyposis, others);
2. Inflammatory bowel disease;
3. Partially excised polyp or endoscopy physician recommending early colonoscopy to document complete excision;
4. Endoscopy physician documenting a rationale for not repeating colonoscopy in future such as co-morbid conditions.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of cases where the colonoscopy physician recommendations matched with the guideline recommendation | 7 months
  % of patients whose recommended colonoscopy frequency is in agreement with guideline recommendation based on patient factors and colonoscopy findings'

SECONDARY OUTCOMES:
Physicians' use of the application (tool reliable) | 7 months
  graded on an ordinal scale (strongly disagree, disagree, neutral, agree, strongly agree), N/A - Have not used app)
Physicians' use of the application (ease of use) | 7 months
  Ease of use graded on an ordinal scale (strongly disagree, disagree, neutral, agree), strongly agree, N/A - Have not used app)
Physicians' use of the application (how familiar is the information in the tool) | 7 months
  graded on an ordinal scale (very familiar, familiar, unsure, new, very new, N/A - Have not used app)
Physicians' use of the application (how often used) | 7 months
  graded on an ordinal scale (every day, every week, every month, less than once a month, did not use it)
Physicians' use of the application (how often used in first month) | 7 months
  graded on an ordinal scale (every day, every week, did not use it)
Physicians' use of the application (how often used during endoscopy slate) | 7 months
  graded on an ordinal scale (never, less than 5%, more than 5% but less than 50%, more than 50%, N/A - have not used the app)
Physicians' use of the application (how often used during non-endoscopy clinical days) | 7 months
  graded on an ordinal scale (never, less than 5%, more than 5% but less than 50%, more than 50%, N/A - have not used the app)
Physicians' use of the application (impact upon decisions) | 7 months
  graded on an ordinal scale (never, less than 5%, more than 5% but less than 50%, more than 50%, N/A - have not used the app)
Physicians' use of the application (likelihood of using tool on ongoing basis in practice) | 7 months
  graded on an ordinal scale (very likely, likely, neutral, not likely, very unlikely )
Physicians' use of the application (main reason provided, among those neutral or unlikely to use on ongoing basis) | 7 months
  graded on an ordinal scale (difficult to use, not helpful, too time consuming, other)
Proportion of cases which have a documented recommendation | 7 months
  % of patients with a documented recommendation

CONTACTS AND LOCATIONS:
Overall Officials: Harminder Singh, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Health Sciences Center, Winnipeg, Manitoba
  - Winnipeg Regional Health Authority, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No
Study findings will be disseminated via presentations at professional forums and published in a peer-reviewed journal.
  No specific feedback will be provided to individual participants as we will perform and report aggregate analysis.

REFERENCES:
- [Background] Potet F, Soullard J. Polyps of the rectum and colon. Gut. 1971 Jun;12(6):468-82. doi: 10.1136/gut.12.6.468. PMID 5314569
- [Background] Muto T, Bussey HJ, Morson BC. The evolution of cancer of the colon and rectum. Cancer. 1975 Dec;36(6):2251-70. doi: 10.1002/cncr.2820360944. PMID 1203876
- [Background] Stryker SJ, Wolff BG, Culp CE, Libbe SD, Ilstrup DM, MacCarty RL. Natural history of untreated colonic polyps. Gastroenterology. 1987 Nov;93(5):1009-13. doi: 10.1016/0016-5085(87)90563-4. PMID 3653628
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Rex DK, Sullivan AW, Perkins AJ, Vemulapalli KC. Colorectal polyp prevalence and aspirational detection targets determined using high definition colonoscopy and a high level detector in 2017. Dig Liver Dis. 2020 Jan;52(1):72-78. doi: 10.1016/j.dld.2019.08.019. Epub 2019 Sep 20. PMID 31543411
- [Background] Leddin D, Lieberman DA, Tse F, Barkun AN, Abou-Setta AM, Marshall JK, Samadder NJ, Singh H, Telford JJ, Tinmouth J, Wilkinson AN, Leontiadis GI. Clinical Practice Guideline on Screening for Colorectal Cancer in Individuals With a Family History of Nonhereditary Colorectal Cancer or Adenoma: The Canadian Association of Gastroenterology Banff Consensus. Gastroenterology. 2018 Nov;155(5):1325-1347.e3. doi: 10.1053/j.gastro.2018.08.017. Epub 2018 Aug 16. PMID 30121253
- [Background] Singh H, Demers AA, Xue L, Turner D, Bernstein CN. Time trends in colon cancer incidence and distribution and lower gastrointestinal endoscopy utilization in Manitoba. Am J Gastroenterol. 2008 May;103(5):1249-56. doi: 10.1111/j.1572-0241.2007.01726.x. Epub 2008 Jan 11. PMID 18190650
- [Background] Lieberman D. How good is your dentist? How good is your endoscopist? The quality imperative. Gastroenterology. 2012 Feb;142(2):194-6. doi: 10.1053/j.gastro.2011.12.016. Epub 2011 Dec 15. No abstract available. PMID 22178380
- [Background] Janssen RM, Takach O, Nap-Hill E, Enns RA. Time to Endoscopy in Patients with Colorectal Cancer: Analysis of Wait-Times. Can J Gastroenterol Hepatol. 2016;2016:8714587. doi: 10.1155/2016/8714587. Epub 2016 Apr 6. PMID 27446872
- [Background] Sey MS, Gregor J, Adams P, Khanna N, Vinden C, Driman D, Chande N. Wait times for diagnostic colonoscopy among outpatients with colorectal cancer: a comparison with Canadian Association of Gastroenterology targets. Can J Gastroenterol. 2012 Dec;26(12):894-6. doi: 10.1155/2012/494797. PMID 23248790
- [Background] Rabeneck L, Paszat LF, Saskin R. Endoscopist specialty is associated with incident colorectal cancer after a negative colonoscopy. Clin Gastroenterol Hepatol. 2010 Mar;8(3):275-9. doi: 10.1016/j.cgh.2009.10.022. Epub 2009 Oct 29. PMID 19879970
- [Background] Pinsky PF, Schoen RE. Contribution of Surveillance Colonoscopy to Colorectal Cancer Prevention. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2937-2944.e1. doi: 10.1016/j.cgh.2020.01.037. Epub 2020 Feb 1. PMID 32017987
- [Background] Leddin D, Enns R, Hilsden R, Fallone CA, Rabeneck L, Sadowski DC, Singh H; Canadian Association of Gastroenterology. Colorectal cancer surveillance after index colonoscopy: guidance from the Canadian Association of Gastroenterology. Can J Gastroenterol. 2013 Apr;27(4):224-8. doi: 10.1155/2013/232769. PMID 23616961
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1131-1153.e5. doi: 10.1053/j.gastro.2019.10.026. Epub 2020 Feb 7. No abstract available. PMID 32044092
- [Background] Rutter MD, East J, Rees CJ, Cripps N, Docherty J, Dolwani S, Kaye PV, Monahan KJ, Novelli MR, Plumb A, Saunders BP, Thomas-Gibson S, Tolan DJM, Whyte S, Bonnington S, Scope A, Wong R, Hibbert B, Marsh J, Moores B, Cross A, Sharp L. British Society of Gastroenterology/Association of Coloproctology of Great Britain and Ireland/Public Health England post-polypectomy and post-colorectal cancer resection surveillance guidelines. Gut. 2020 Feb;69(2):201-223. doi: 10.1136/gutjnl-2019-319858. Epub 2019 Nov 27. PMID 31776230
- [Background] Saini SD, Nayak RS, Kuhn L, Schoenfeld P. Why don't gastroenterologists follow colon polyp surveillance guidelines?: results of a national survey. J Clin Gastroenterol. 2009 Jul;43(6):554-8. doi: 10.1097/MCG.0b013e31818242ad. PMID 19542818
- [Background] Menees SB, Elliott E, Govani S, Anastassiades C, Schoenfeld P. Adherence to recommended intervals for surveillance colonoscopy in average-risk patients with 1 to 2 small (<1 cm) polyps on screening colonoscopy. Gastrointest Endosc. 2014 Apr;79(4):551-7. doi: 10.1016/j.gie.2014.01.029. PMID 24630082
- [Background] van Heijningen EM, Lansdorp-Vogelaar I, Steyerberg EW, Goede SL, Dekker E, Lesterhuis W, ter Borg F, Vecht J, Spoelstra P, Engels L, Bolwerk CJ, Timmer R, Kleibeuker JH, Koornstra JJ, de Koning HJ, Kuipers EJ, van Ballegooijen M. Adherence to surveillance guidelines after removal of colorectal adenomas: a large, community-based study. Gut. 2015 Oct;64(10):1584-92. doi: 10.1136/gutjnl-2013-306453. Epub 2015 Jan 13. PMID 25586057
- [Background] Hong S, Suh M, Choi KS, Park B, Cha JM, Kim HS, Jun JK, Han DS. Guideline Adherence to Colonoscopic Surveillance Intervals after Polypectomy in Korea: Results from a Nationwide Survey. Gut Liver. 2018 Jul 15;12(4):426-432. doi: 10.5009/gnl17403. PMID 29429156
- [Background] Djinbachian R, Dube AJ, Durand M, Camara LR, Panzini B, Bouchard S, von Renteln D. Adherence to post-polypectomy surveillance guidelines: a systematic review and meta-analysis. Endoscopy. 2019 Jul;51(7):673-683. doi: 10.1055/a-0865-2082. Epub 2019 Mar 25. PMID 30909308
- [Background] Kahi CJ, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Lieberman D, Levin TR, Robertson DJ, Rex DK; United States Multi-Society Task Force on Colorectal Cancer. Colonoscopy Surveillance After Colorectal Cancer Resection: Recommendations of the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2016 Mar;150(3):758-768.e11. doi: 10.1053/j.gastro.2016.01.001. Epub 2016 Feb 10. PMID 26892199
- [Background] Singh H, Kaita L, Taylor G, Nugent Z, Bernstein C. Practice and documentation of performance of colonoscopy in a central Canadian health region. Can J Gastroenterol Hepatol. 2014 Apr;28(4):185-90. doi: 10.1155/2014/635932. PMID 24729991
- [Background] Read AJ, Weissman A, Schoenfeld PS, Saini S, Menees SB, Saini SD. Who is Responsible for What Happens Before, During, and After Colonoscopy? Results of a National Survey of Primary Care Physicians. J Clin Gastroenterol. 2018 Jul;52(6):e44-e47. doi: 10.1097/MCG.0000000000000881. PMID 28737648
- [Background] Leddin D, Hunt R, Champion M, Cockeram A, Flook N, Gould M, Kim YI, Love J, Morgan D, Natsheh S, Sadowski D; Canadian Association of Gastroenterology; Canadian Digestive Health Foundation. Canadian Association of Gastroenterology and the Canadian Digestive Health Foundation: Guidelines on colon cancer screening. Can J Gastroenterol. 2004 Feb;18(2):93-9. doi: 10.1155/2004/983459. No abstract available. PMID 14997217
- [Background] Leddin DJ, Enns R, Hilsden R, Plourde V, Rabeneck L, Sadowski DC, Signh H. Canadian Association of Gastroenterology position statement on screening individuals at average risk for developing colorectal cancer: 2010. Can J Gastroenterol. 2010 Dec;24(12):705-14. doi: 10.1155/2010/683171. PMID 21165377
- [Background] Rex DK, Ahnen DJ, Baron JA, Batts KP, Burke CA, Burt RW, Goldblum JR, Guillem JG, Kahi CJ, Kalady MF, O'Brien MJ, Odze RD, Ogino S, Parry S, Snover DC, Torlakovic EE, Wise PE, Young J, Church J. Serrated lesions of the colorectum: review and recommendations from an expert panel. Am J Gastroenterol. 2012 Sep;107(9):1315-29; quiz 1314, 1330. doi: 10.1038/ajg.2012.161. Epub 2012 Jun 19. PMID 22710576
- [Background] Donner A, Klar N. Design and analysis of cluster randomization trials in health research. New York. 2010.
- [Background] Elias ED, Targownik LE, Singh H, Bernstein CN. A Population-Based Study of Combination vs Monotherapy of Anti-TNF in Persons With IBD. Inflamm Bowel Dis. 2020 Jan 1;26(1):150-157. doi: 10.1093/ibd/izz148. PMID 31340002
- [Background] Austin PC. A comparison of the statistical power of different methods for the analysis of cluster randomization trials with binary outcomes. Stat Med. 2007 Aug 30;26(19):3550-65. doi: 10.1002/sim.2813. PMID 17238238
- [Background] Rotondi M. Sample size estimation functions for cluster randomized trials (Version 1.0)[Software]. Retrieved December. 2015;8:2017.
- [Background] Parker DR, Evangelou E, Eaton CB. Intraclass correlation coefficients for cluster randomized trials in primary care: the cholesterol education and research trial (CEART). Contemp Clin Trials. 2005 Apr;26(2):260-7. doi: 10.1016/j.cct.2005.01.002. PMID 15837446
- [Background] Kul S, Vanhaecht K, Panella M. Intraclass correlation coefficients for cluster randomized trials in care pathways and usual care: hospital treatment for heart failure. BMC Health Serv Res. 2014 Feb 24;14:84. doi: 10.1186/1472-6963-14-84. PMID 24565441
- [Background] Elley CR, Kerse N, Chondros P, Robinson E. Intraclass correlation coefficients from three cluster randomised controlled trials in primary and residential health care. Aust N Z J Public Health. 2005 Oct;29(5):461-7. doi: 10.1111/j.1467-842x.2005.tb00227.x. PMID 16255449
- [Derived] Shaffer SR, Lambert P, Unruh C, Harland E, Helewa RM, Decker K, Singh H. Optimizing Timing of Follow-Up Colonoscopy: A Pilot Cluster Randomized Trial of a Knowledge Translation Tool. Am J Gastroenterol. 2024 Mar 1;119(3):547-555. doi: 10.14309/ajg.0000000000002542. Epub 2023 Oct 3. PMID 37787644